CLINICAL TRIAL: NCT01590004
Title: Technical Description of Cooled Radiofrequency Ablation of Lumbar Medial Branches for the Treatment of Lumbar Facet Pain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mehul Desai (Industry)
Collaborators: Halyard Health (Industry)
Responsible Party: Sponsor-Investigator, Mehul Desai, Principal Investigator, MAPS Applied Research Center
Organization: MAPS Applied Research Center (Industry)
Other Study IDs: lumbar01
Record Dates: First submitted 2012-04-30; First posted 2012-05-02 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Lumbar Facet Joint Pain
Keywords: LumbarCool system; Cooled radiofrequency medial ablation; Cooled-RF neurotomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study aims to develop a technical description of lumbar medial branch ablation using the LumbarCool system. The procedure uses cooled radiofrequency (cooled-RF) technology in treating patients with diagnosed lumbar facet joint pain.

DETAILED DESCRIPTION:
This is a prospective, open-label, single center clinical study to be enrolled at George Washington University Medical Center. This study will consist of 10 patients and each patient will be assessed at pre-treatment, pre-discharge, and at 1 and 3 months post treatment. Outcomes to be evaluated include: pain severity, disability, and the occurrence of adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Literate
2. Aged between 18 and 75 years
3. Chronic lumbar pain for > 6 months
4. 3-day average NRS score at least 4 and not greater than 8
5. Clinical features consistent with possible lumbar z-joint pain (such as pain and tenderness over not more than three segments unilaterally)
6. No adequate relief with conservative management, including physical therapy, chiropractic manipulation, exercises, and drug therapy
7. Understand and tolerate lumbar medial branch diagnostic blocks
8. Positive for lumbar zygapophyseal joint pain after comparative diagnostic blocks (≥ 80% pain relief) per standard of care.
9. Understands study protocol and provides voluntary written consent to participate in study and outcome measurements
10. Normal neurological exam
11. Understands and agrees to use an acceptable form of birth control

Exclusion Criteria:

1. Current pregnancy, currently breast feeding or the intent of becoming pregnant during the study period
2. Prior posterior lumbar fusion
3. Prior low back surgery
4. Concurrent cervical or thoracic pain or pain in these regions lasting longer than 2 weeks during the last 6 months
5. Compensable disability or work injury or ongoing litigation
6. Prior treatment with radiofrequency neurotomy in the lumbar region within 3 months
7. Discogenic pain verified by controlled discography
8. Sources of pain not in the lumbar spine
9. Leg pain greater than back pain
10. Obvious inappropriate pain behavior during physical exam
11. Neurologic deficits
12. Positive straight leg raising result
13. Any features of upper motor neuron lesion
14. Gait abnormality not attributable to spinal pain
15. Severe Central Spinal Canal Stenosis (> 50%) evident on prior computed tomogram or magnetic resonance image
16. Spondylolysis
17. Spondylolisthesis
18. More than 75% narrowing of a disc space on plain radiographs
19. Spondyloarthropathy
20. Score higher than 20 on the Beck Depression Inventory
21. Patients addicted to alcohol, narcotics or other illegal substances
22. Dependence on opioids
23. Uncontrolled acute/chronic illness that may confound interpretation of outcome measures
24. Allergy to injectants, medication or anesthetics to be used
25. Active or uncontrolled rheumatoid arthritis or other autoimmune diseases
26. Patients with a history of mental instability or diagnosed with a mental disorder
27. Patient unwilling or unable to comply with study procedures or follow-up visits
28. The presence of a pacemaker in the patient

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of Medical Advanced Pain Specialists, PA (MAPS)
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2012-08; Primary Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Confirm acute safety of the procedure | Baseline to 3 months post procedure.
  The primary outcome is to confirm acute safety of the procedure utilizing the neurological exam.
  The following outcome measures will also be used to confirm there are no safety concerns at one month and 3 months follow-up visits:
  * Pain intensity using the Numerical Rating Scale (NRS)
  * Change in medication usage
  * Assessment of adverse device effects, including neurological exam (light touch/pin prick, strength, straight leg test, gait, heel to toe/straight-line walking, heel to shin) (immediately post procedure, 1 month and 3 months).

CONTACTS AND LOCATIONS:
Overall Officials: Mehul J Desai, MD, Principal Investigator — MAPS Applied Research Center
Locations (1):
- MAPS Applied Research Center, Inc., Edina, Minnesota, United States